CLINICAL TRIAL: NCT04128150
Title: High Resolution Retina Imaging
Acronym: IHR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A03223-50; 2017-A03223-50 (Other: N° IDRCB)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Retinitis Pigmentosa; Maculopathy, Age Related; Macular Dystrophy; Macular Edema; Retinal Degeneration; Diabetic Retinopathy; Occlusion Retinal Vein; Hypertension
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration; Macular Edema; Retinal Degeneration; Diabetic Retinopathy; Retinal Vein Occlusion; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To increase the clinical experience of using the rtx1 camera in various retinal disorders and to follow the evolution of structural alterations during retinal diseases using adaptive optics imaging with the rtx1 camera

ELIGIBILITY:
Inclusion Criteria:

* Persons over 12 years of age, of both sexes, presenting with retinal pathologies.
* Beneficiaries of the health insurance

Exclusion Criteria:

* Any abnormality preventing good quality OA imaging on both eyes
* Major under guardianship or curatorship

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathologies affecting photoreceptors and the retinal vessels
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of retina diseases | From date of inclusion until the date of last documented progression , assessed up to 5 years
  Increase the clinical experience of using the rtx1 camera in various conditions with retinal impact

CONTACTS AND LOCATIONS:
Overall Officials: Michel PAQUES, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vints
Locations (3):
- France (3):
  - Hôpital Lariboisière, Paris
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - Hôpital Pitié-Salpétrière, Paris

REFERENCES:
- [Derived] Paques M, Norberg N, Chaumette C, Sennlaub F, Rossi E, Borella Y, Grieve K. Long Term Time-Lapse Imaging of Geographic Atrophy: A Pilot Study. Front Med (Lausanne). 2022 Jun 22;9:868163. doi: 10.3389/fmed.2022.868163. eCollection 2022. PMID 35814763